CLINICAL TRIAL: NCT02704832
Title: Role of Geriatric Intervention in Treatment of Older Patients With Cancer : a Phase III Randomized Study (PREPARE)
Brief Title: Role of Geriatric Intervention in Treatment of Older Patients With Cancer (PREPARE)
Acronym: PREPARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IB 2015-08; ID-RCB number 2015-A01417-42 (Other: ANSM)
Record Dates: First submitted 2016-02-19; First posted 2016-03-10 (Estimated); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Colorectal Cancer; Lung Cancer; Prostate Cancer; Bladder Cancer; Ovarian Cancer; Lymphoma
Keywords: Geriatric oncology; Intervention; Case management
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Urinary Bladder Neoplasms; Ovarian Neoplasms; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (No Intervention): Arm A "Standard oncological care": patients will be treated according to daily oncological practices as defined for each type of cancer, in the "Management protocol of Oncology" written and validated by a group of expert oncologists. The quality of life will be assessed every 3 months during the first year and at 18 months. The study's follow-up will last until 3 years after the enrollment of the last patient and data on vital status of the patient, weight, place of life and the status of the disease will be collected every 6 months.
- Arm B (Experimental): Arm B "Geriatrician Intervention": patients will be treated according to the same "Management protocol of Oncology" than patients in the arm "Standard oncological care".
  * Before the beginning of the medical treatment, a comprehensive geriatric assessment will be performed by the geriatrician and the nurse that will define a plan of geriatric management care, according to the "Management protocol of Geriatrics".
  * The nurse, under the supervision of a geriatrician, will monitor implemented geriatric interventions. Phone follow-up will be performed every month for 6 months and at 9 months or during any change of situation according to a pre-established phone call plan. A full geriatric assessment by the geriatrician and the nurse will be performed at 6 and 12 months.
  Interventions: Other: Geriatrician Intervention

INTERVENTIONS:
Other: Geriatrician Intervention — Arm B : The duration of the geriatric intervention will be 12 months. The quality of life will be assessed every 3 months during the first year and at 18 months. The study's follow-up will last until 3 years after the enrollment of the last patient and data on vital status of the patient, weight, place of life and the status of the disease will be collected every 6 months.
  Arms: Arm B

SUMMARY:
Randomized trials have already demonstrated that geriatric intervention was able to improve survival in the general elderly population but only a few have been performed in cancer patients. At the end, these data are not sufficient to consider geriatric intervention as validated in this setting. Case Management, coordinated by a geriatrician and a trained nurse, could improve prognosis of elderly patients with cancer. This approach, can be integrated in daily oncology practice. This strategy will be compared to usual oncological management in a randomized phase III trial.

DETAILED DESCRIPTION:
Patients will first be screened using the G8 screening tool. If the resulting score is altered (G8 <= 14), patients will be included in the main study and randomized according to 2 modalities: Arm A / Usual care (treatment according to on-going regimens in oncology) or Arm B /Case management (assessment of the patient by the nurse and the geriatrician with interventions as prescribed by the geriatrician). The intervention will be considered effective if, at one year, compared to usual care there is a significant clinical improvement in overall survival (OS) without a significant deterioration or/and clinical improvement of at least one of the targeted quality of life (QoL) scores, without significant clinical deterioration in at least one of the targeted QoL scores and without significant difference in OS in favor of usual care.

If the resulting score is normal (G8 > 14), patients will be treated according to their physician-in-charge opinion. A minimal set of data will be collected (age, sex, tumor type, disease stage, performance status (PS), creatinine clearance, albumin and C-Reactive Protein (CRP) levels mainly) to allow for the characterization of the population in order to compare our results to those of other published series.

ELIGIBILITY:
Inclusion Criteria:

1. Patient older 70 years and older
2. Performance status 0 to 3 (WHO)
3. G8 and QLQ-C30 questionnaires 'score are available
4. No previous geriatric evaluation during cancer treatment
5. Locally advanced or metastatic disease :

   1. 1st line medical treatment :

      * Breast cancer : locally advanced or metastatic disease, hormone-resistant and Her2 negative,
      * Colon and rectum : metastatic (unresectable metastasis),
      * Prostate cancer : metastatic and refractory to hormonal castration,
      * Bladder cancer : locally advanced or metastatic,
      * Ovarian cancer : advanced stage (IIb to IV),
      * Lung cancer : metastatic non-small cell,
      * Lymphomas (indolent and aggressive)
   2. Or 2nd line medical treatment :

      * Breast cancer : locally advanced or metastatic disease, hormone-resistant and Her2 negative,
      * Colon and rectum : metastatic (unresectable metastasis),
      * Prostate cancer : metastatic and refractory to hormonal castration,
      * Ovarian cancer : advanced stage (IIb to IV),
      * Lymphomas (indolent and aggressive)
6. Life expectancy over 6 months
7. Signed informed consent
8. Patients with a French social security in compliance with the French law relating to biomedical research (Article L.1121-11 of French Public Health Code).

Exclusion Criteria:

1. Patient who already received 2 medical treatment lines
2. Exclusive 1st or 2nd treatment lines of :

   * Hormonotherapy (except for prostate cancer : abiteratone acetate is allowed),
   * Surgery,
   * Radiotherapy,
3. "Best supportive care" treatment
4. Patient unable to understand quality of life questionnaire
5. Patient unable to follow and comply with the study procedures because of any geographical, social or psychological reasons.
6. Patient placed under guardianship
7. Planned concomitant participation to another medical interventional trial during the 12 months following the inclusion in the randomized study PREPARE
8. Previous enrolment in the present study

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 792 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-11-21 (Actual)

PRIMARY OUTCOMES:
Overall survival defined as the delay between randomization and death, all causes. | Year 1
Health related quality of life (HR-QoL) assessed using 3 scales of European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaire. | Year 1

SECONDARY OUTCOMES:
Overall survival defined as the delay between randomization and death, all causes. | Year 3
Health related quality of life (hRQoL) assessed using 3 scales of EORTC QLQ-C30 questionnaire. | Year 3
6-month response rates defined as per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 or Cheson criteria. | Month 6
Toxicity graded according to National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4. | up to 3 years
Number of unscheduled hospitalizations. | up to 3 years
Length of unscheduled hospitalizations. | up to 3 years
For the experimental arm only: Assessment of autonomy using Activities of Daily Living (ADL) questionnaire. | Months 0, 6, 12
For the experimental arm only: Assessment of autonomy using Instrumental Activities of Daily Living (IADL) questionnaire. | Months 0, 6, 12
For the experimental arm only: Assessment of depression using Geriatric Depression Scale (GDS-15) scale. | Months 0, 6, 12
For the experimental arm only: Assessment of cognitive functions using mini mental state exam (MMSE). | Months 0, 6, 12
For the experimental arm only: Assessment of comorbidities using Cumulative Illness Rating Scale for Geriatrics (CIRS-G) scale. | Months 0, 6, 12
For the experimental arm only: Assessment of nutritional status using mini nutritional assessment (MNA) scale. | Months 0, 6, 12
For the experimental arm only: Assessment of mobility using get-up and Go test. | Months 0, 6, 12

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Louis SOUBEYRAN, PU-PH, Study Chair — Institut Bergonié
Locations (50):
- France (50):
  - Centre Hospitalier Universitaire de Grenoble, Grenoble, Auvergne-Rhône-Alpes
  - Institut de Cancérologie de l'Ouest, Angers
  - Centre Hospitalier de Beauvais, Beauvais
  - Clinique Anne d'Artois, Béthune
  - Institut Bergonié Centre Régional de Lutte Contre le Cancer, Bordeaux
  - CHU de Bordeaux, Bordeaux
  - Centre Hospitalier Universitaire de Caen, Caen
  - Infirmerie Protestante de Lyon, Caluire-et-Cuire
  - Centre Hospitalier Intercommunal de Castres Mazamet, Castres
  - Centre Hospitalier Métropôle Savoie Chambéry, Chambéry
  - Centre Hospitalier de Chinon, Chinon
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - Centre Jean Perrin, Clermont-Ferrand
  - AP-HP Henri Mondor, Créteil
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Hospitalier de Dax, Dax
  - Centre Georges François Leclerc, Dijon
  - Centre Hospitalier Universitaire de Martinique, Fort de France
  - Centre Hospitalier Emile Roux, Le Puy-en-Velay
  - Centre Hospitalier Universitaire de Lille, Lille
  - Clinique Mutualiste Eugène André, Lyon
  - Hôpital Saint Joseph Saint Luc, Lyon
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Hospitalier de Mont de Marsan, Mont-de-Marsan
  - Institut de Cancérologie de Montpellier, Montpellier
  - Institut de Cancérologie de Lorraine, Nancy
  - Centre Catherine de Sienne, Nantes
  - Centre Hospitalier Universitaire de Nîmes, Nîmes
  - AP-HP Hôpital Saint Louis, Paris
  - Centre Hospitalier de Pau, Pau
  - Polyclinique Francheville, Périgueux
  - Hospices Civils de Lyon, Pierre-Bénite
  - Centre CARIO - HPCA, Pleurin Sur Mer
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Centre Hospitalier René Dubos, Pontoise
  - Centre Hospitalier Annecy Genevois, Pringy
  - Centre Hospitalier Intercommunal de Cornouaille, Quimper
  - Centre Jean Godinot, Reims
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - Centre Eugène Marquis, Rennes
  - Centre Hospitalier Universitaire de Rouen, Rouen
  - Centre Hospitalier Privé de Saint Grégoire, Saint-Grégoire
  - Centre Hospitalier Universitaire de Nantes, Saint-Herblain
  - GHPSO Senlis Creil Picardie, Senlis
  - Centre Hospitalier de Saint-Malo, St-Malo
  - Centre Hospitalier Universitaire de Strasbourg, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Centre Hospitalier de Tourcoing, Tourcoing
  - Centre Hospitalier Universitaire de Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Soubeyran P, Terret C, Bellera C, Bonnetain F, Jean OS, Galvin A, Chakiba C, Zwolakowski MD, Mathoulin-Pelissier S, Rainfray M. Role of geriatric intervention in the treatment of older patients with cancer: rationale and design of a phase III multicenter trial. BMC Cancer. 2016 Dec 1;16(1):932. doi: 10.1186/s12885-016-2927-4. PMID 27908282